CLINICAL TRIAL: NCT05808998
Title: A Clinical Trial of Stereotactic Radiotherapy on Spinal Metastasis
Brief Title: A Single-center Observational Clinical Trial of Stereotactic Radiotherapy on Metastatic Spinal Tumors Using TomoTherapy
Acronym: SM-SBRT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-SM-SBRT
Record Dates: First submitted 2023-03-11; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Spinal Bone Metastases; Radiation Therapy
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Stereotactic body radiotherapy using TomoTherapy

SUMMARY:
A single-center observational clinical trial will be performed for metastatic spinal tumors by stereotactic radiotherapy using TomoTherapy. In this study, we will explore the local control rate (LCR), disease-free progression time (PFS), overall survival time (OS), and pain relief in patients with spinal metastasis, so as to provide a basis for developing relevant guidelines or consensus.

DETAILED DESCRIPTION:
In this observational single-arm study, a total of 45 patients with metastatic spinal tumors will be enrolled. The patients were aged between 18 and 75 years old. And all the subjects should meet the inclusion criteria and sign the informed consent. Meanwhile, the patients' medical history characteristics, including gender, age, imaging data (X-ray, CT, MRI, or PET-CT, etc.), primary tumor type, pathological type, previous treatment, previous disease history, tumor markers and bone metabolism indexes were collected and recorded on the CRF. The metastatic spinal tumors by stereotactic radiotherapy(SBRT) using TomoTherapy. The adiotherapy dose is 6Gy×5Fx, 5Gy×5Fx or 4Gy×5Fx according to the irradiation site. Treatment should be interrupted if there is severe bone marrow suppression, vertebral compression fracture, or radiation myelitis. The adjacentnormal tissue constrains refer to the UK SABR Consortium Guidelines (2022 version). Follow-up was performed 1 month after radiotherapy, thereafter every 3 months for 1-4 years. The parameters includ blood routine, liver and kidney function, bleeding and coagulation function, bone metabolism index, tumor markers, bone metastasis imaging examination. Tumor response will refer to the Cancer Response Criteria and Bone Metastases: RECIST 1.1, MDA and PERCIST.

ELIGIBILITY:
Inclusion Criteria:

1. Spinal metastasis diagnosed by emission computed tomography, X-ray examination, computed tomography, magnetic resonance imaging (MRI) or 18F-fluorodeoxy glucose positron emission tomography within 6 weeks before enrollment;
2. Patients with unresectable spinal metastases;
3. SBRT was for patients with painful spinal metastases, physiological hypofunction, decreased behavioral capacity and quality of life. And SBRT was used to help to prevent or delay skeletal related event (SRE). Including postoperative radiotherapy (especially post-separation), single or salvage radiotherapy;
4. age 18-75 years old;
5. KPS score equal to 70 points or over;
6. Patients were required to have histologically confirmed metastatic disease from solid tumors, such as breast cancer, renal carcinoma or liver cancer;
7. The distance between metastatic lesion and spinal cord was more than 3mm；
8. Hemoglobin >90g/L, white cells count≥3.5×109/L, platelet count≥80×109/L, within 1 week before treatment;
9. No birth plans for the duration of study participation and up to 3 months following completion of therapy;
10. Sign the informed consent.

Exclusion Criteria:

1. Spinal cord or cauda equina compression, the rapid decrement of neurological function or paralysis;
2. A compression fracture of the spine, spinal instability and subsequent inability to lie on back;
3. Metastatic lesions more than 5cm;
4. Multilevel segments involvement, including more than 5 metastatic segments, or 3 isolated lesions, or exceed two adjacent vertebrae;
5. The treatment site had received prior radiotherapy prior to the initiation of the study;
6. Complicated with other malignant tumors or severe internal diseases affected the prognosis;
7. Cannot tolerate radiation therapy, including the ones with scleroderma or connective tissue diseases, or cann't complete the radiation treatment according to the research;
8. Pregnant women or breast feeding mothers;
9. Systemic radionuclide therapy within 30 days before SBRT, or external radiotherapy within 90 days before SBRT;
10. Pathologically confirmed as myeloma or lymphoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 45 patients with spinal metastases were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
1-year local control rate | 2024.4-2025.4
  The proportion of complete remission, partial remission, stable disease, and disease progression patients in the total number of enrolled cases. Tumor response will refer to the Cancer Response Criteria and Bone Metastases: RECIST 1.1, MDA and PERCIST.

SECONDARY OUTCOMES:
1- and 2- year overall survival (OS) | 2024.4-2026.4
  year overall survival (OS): From day of radiotherapy until the date of death or the end in 1 year, 2-year OS: From day of radiotherapy until the date of death or the end in 2 years
1- and 2-year Progression-Free Survival(PFS) | 2024.4-2026.4
  1-year Progression-Free Survival (PFS)：From day of radiotherapy until the Progression of bone metastases sites in 1 year, 2-year PFS：From day of radiotherapy until the Progression of bone metastases sites in 2 years
Pain relief | 2024.4-2026.4
  Assessment of pain will be according to the Numerical Rating Scale (NRS).
Bone metastasis-related events (SRE) | 2024.4-2026.4
  Bone metastasis-related events will be recorded, including pathological fracture and spinal cord compression, etc.
Epidural spinal cord compression (ESCC) grade | 2024.4-2026.4
  Epidural spinal cord compression (ESCC) grade will be assessed refer to ESCC scale.
Adverse reactions | 2024.4-2026.4
  1-Number of participants with treatment-related adverse events as assessed by CTCAE v4.0.